CLINICAL TRIAL: NCT01154816
Title: A Phase II Study of MLN8237, a Selective Aurora A Kinase Inhibitor in Children With Recurrent/Refractory Solid Tumors and Leukemias
Brief Title: Alisertib in Treating Young Patients With Recurrent or Refractory Solid Tumors or Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ADVL0921; NCI-2011-02051 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000680512; ADVL0921 (Other: Childrens Oncology Group); ADVL0921 (Other: CTEP); U10CA098543 (NIH)
Record Dates: First submitted 2010-06-30; First posted 2010-07-01 (Estimated); Results first posted 2017-06-05 (Actual); Last update posted 2020-05-13 (Actual); Status verified 2017-09

CONDITIONS: Hepatoblastoma; Previously Treated Childhood Rhabdomyosarcoma; Recurrent Childhood Acute Lymphoblastic Leukemia; Recurrent Childhood Acute Myeloid Leukemia; Recurrent Childhood Kidney Neoplasm; Recurrent Childhood Malignant Germ Cell Tumor; Recurrent Childhood Rhabdomyosarcoma; Recurrent Childhood Soft Tissue Sarcoma; Recurrent Ewing Sarcoma/Peripheral Primitive Neuroectodermal Tumor; Recurrent Neuroblastoma; Recurrent Osteosarcoma
MeSH Terms: conditions — Hepatoblastoma; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Neuroectodermal Tumors, Primitive, Peripheral; Neuroblastoma; Osteosarcoma | interventions — MLN 8237

ARMS (12):
- Arm I (neuroblastoma- measurable) (Experimental): Patients with measurable neuroblastoma receive alisertib PO QD on days 1-7. Treatment repeats every 21 days for up to 35 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Alisertib; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study
- Arm II (Neuroblastoma- MIBG evaluable) (Experimental): Patients MIBG evaluable neuroblastoma receive alisertib PO QD on days 1-7. Treatment repeats every 21 days for up to 35 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Alisertib; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study
- Arm III (rhabdomyosarcoma) (Experimental): Patients with rhabdomyosarcoma receive alisertib PO QD on days 1-7. Treatment repeats every 21 days for up to 35 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Alisertib; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study
- Arm IV (osteosarcoma) (Experimental): Patients with osteosarcoma receive alisertib PO QD on days 1-7. Treatment repeats every 21 days for up to 35 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Alisertib; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study
- Arm V (Ewing sarcoma/peripheral PNET) (Experimental): Patients with Ewing sarcoma/peripheral PNET receive alisertib PO QD on days 1-7. Treatment repeats every 21 days for up to 35 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Alisertib; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study
- Arm VI (non-RMS soft tissue sarcoma) (Experimental): Patients with non-RMS soft tissue sarcoma receive alisertib PO QD on days 1-7. Treatment repeats every 21 days for up to 35 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Alisertib; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study
- Arm VII (hepatoblastoma) (Experimental): Patients hepatoblastoma receive alisertib PO QD on days 1-7. Treatment repeats every 21 days for up to 35 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Alisertib; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study
- Arm VIII (malignant germ cell tumor) (Experimental): Patients with malignant germ cell tumor receive alisertib PO QD on days 1-7. Treatment repeats every 21 days for up to 35 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Alisertib; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study
- Arm IX (Wilms tumor) (Experimental): Patients with Wilms tumor receive alisertib PO QD on days 1-7. Treatment repeats every 21 days for up to 35 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Alisertib; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study
- Arm X (acute lymphoblastic leukemia) (Experimental): Patients with acute lymphoblastic leukemia receive alisertib PO QD on days 1-7. Treatment repeats every 21 days for up to 35 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Alisertib; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study
- Arm XI (acute myelogenous leukemia) (Experimental): Patients acute myelogenous leukemia receive alisertib PO QD on days 1-7. Treatment repeats every 21 days for up to 35 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Alisertib; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study
- Arm XII (rhabdoid malignancy) (Experimental): Patients with rhabdoid malignancy receive alisertib PO QD on days 1-7. Treatment repeats every 21 days for up to 35 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Alisertib; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study

INTERVENTIONS:
Drug: Alisertib — Given orally
  Other Names: Aurora A Kinase Inhibitor MLN8237; MLN-8237; MLN8237
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Pharmacological Study — Correlative studies

SUMMARY:
This phase II trial is studying the side effects of and how well alisertib works in treating young patients with relapsed or refractory solid tumors or leukemia. Alisertib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the objective response rate to MLN8237 (alisertib) in children with relapsed or refractory solid tumors and leukemias, administered once daily for 7 days every 21 days.

SECONDARY OBJECTIVES:

I. To further define and describe the toxicities of MLN8237 administered on this schedule.

II. To further characterize the pharmacokinetics of MLN8237 in children with refractory cancer.

III. To evaluate aurora A kinase expression using immunohistochemistry in solid tumors and leukemic blasts from tissue obtained at diagnosis and, if available, at relapse.

IV. To explore the relationship between polymorphic variations in the UDP-glucuronosyltransferase gene UGT1A1 and exposure to MLN8237, and to assess 2 common polymorphic variants in the aurora A kinase gene, Phe31Ile and Val57Ile.

OUTLINE: This is a multicenter study. Patients are stratified according to type of tumor (measurable neuroblastoma vs neuroblastoma with metaiodobenzylguanidine [MIBG]-positive lesions vs osteosarcoma vs Ewing sarcoma/primitive neuroectodermal tumor [PNET] vs rhabdosarcoma vs non-rhabdomyosarcoma [RMS] soft tissue sarcoma vs hepatoblastoma vs malignant germ cell tumor vs Wilms tumor vs acute myeloid leukemia [AML] vs acute lymphoblastic leukemia [ALL] vs rhabdoid tumors).

ARM I (NEUROBLASTOMA- MEASURABLE): Patients receive alisertib orally (PO) once daily (QD) on days 1-7. Treatment repeats every 21 days for up to 35 courses in the absence of disease progression or unacceptable toxicity.

ARM II (NEUROBLASTOMA-MIBG EVALUABLE): Patients receive alisertib PO QD on days 1-7. Treatment repeats every 21 days for up to 35 courses in the absence of disease progression or unacceptable toxicity.

ARM III (RHABDOMYOSARCOMA): Patients receive alisertib PO QD on days 1-7. Treatment repeats every 21 days for up to 35 courses in the absence of disease progression or unacceptable toxicity.

ARM IV (OSTEOSARCOMA): Patients receive alisertib PO QD on days 1-7. Treatment repeats every 21 days for up to 35 courses in the absence of disease progression or unacceptable toxicity.

ARM V (EWING SARCOMA/ PERIPHERAL PNET): Patients receive alisertib PO QD on days 1-7. Treatment repeats every 21 days for up to 35 courses in the absence of disease progression or unacceptable toxicity.

ARM VI (NON-RMS SOFT TISSUE SARCOMA): Patients receive alisertib PO QD on days 1-7. Treatment repeats every 21 days for up to 35 courses in the absence of disease progression or unacceptable toxicity.

ARM VII (HEPATOBLASTOMA): Patients receive alisertib PO QD on days 1-7. Treatment repeats every 21 days for up to 35 courses in the absence of disease progression or unacceptable toxicity.

ARM VIII (MALIGNANT GERM CELL TUMOR): Patients receive alisertib PO QD on days 1-7. Treatment repeats every 21 days for up to 35 courses in the absence of disease progression or unacceptable toxicity.

ARM IX (WILMS TUMOR): Patients receive alisertib PO QD on days 1-7. Treatment repeats every 21 days for up to 35 courses in the absence of disease progression or unacceptable toxicity.

ARM X (ACUTE LYMPHOBLASTIC LEUKEMIA): Patients receive alisertib PO QD on days 1-7. Treatment repeats every 21 days for up to 35 courses in the absence of disease progression or unacceptable toxicity.

ARM XI (ACUTE MYELOGENOUS LEUKEMIA): Patients receive alisertib PO QD on days 1-7. Treatment repeats every 21 days for up to 35 courses in the absence of disease progression or unacceptable toxicity.

ARM XII (RHABDOID MALIGNANCY): Patients receive alisertib PO QD on days 1-7. Treatment repeats every 21 days for up to 35 courses in the absence of disease progression or unacceptable toxicity.

Plasma samples are collected from all patients at baseline and periodically during course 1 for pharmacokinetic and other studies.

After completion of study therapy, patients are followed up for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have had histologic verification of malignancy at original diagnosis or at relapse, to include any of the following malignancies (no other histology is eligible):

  * Neuroblastoma- measurable
  * Neuroblastoma- MIBG evaluable
  * Rhabdomyosarcoma
  * Osteosarcoma
  * Ewing sarcoma/Peripheral PNET
  * Non-RMS soft tissue sarcoma
  * Hepatoblastoma
  * Malignant germ cell tumor
  * Wilms tumor
  * Acute lymphoblastic leukemia
  * Acute myelogenous leukemia
  * Rhabdoid malignancy
* Disease status for solid tumor patients:

  * Patients must have radiographically measurable disease (with the exception of neuroblastoma)
  * Measurable disease is defined as the presence of at least one lesion on magnetic resonance imaging (MRI) or computed tomography (CT) scan that can be accurately measured with the longest diameter a minimum of 20 mm in at least one dimension; for spiral CT, measurable disease is defined as a minimum diameter of 10 mm in at least one dimension
  * Note: The following do not qualify as measurable disease:

    * Malignant fluid collections (e.g., ascites, pleural effusions)
    * Bone marrow infiltration
    * Lesions detected by nuclear medicine studies (e.g., bone, gallium or positron emission tomography [PET] scans)
    * Elevated tumor markers in plasma or cerebrospinal fluid (CSF)
    * Previously irradiated lesions that have not demonstrated clear progression post radiation
  * Patients with neuroblastoma who do not have measurable disease but have MIBG+ evaluable disease are eligible
* Disease status for leukemia patients:

  * Patients with leukemia must be recurrent or refractory to at least two prior induction or treatment regimens, in addition to the following criteria:
  * Acute lymphoid leukemia:

    * 25% blasts in the bone marrow (M3 bone marrow), excluding patients with known central nervous system (CNS) disease
  * Acute myeloid leukemia according to FAB classification

    * ≥ 5 % blasts in the bone marrow (M2/M3 bone marrow); excluding patients with known CNS disease
* Rhabdoid tumors:

  * To be eligible for enrollment in the rhabdoid tumors stratum, the patient must have a solid tumor where the institutional pathological evaluation of the tumor at initial diagnosis or relapse has confirmed:

    * Morphology and immunophenotypic panel consistent with rhabdoid tumor (required)
    * Loss of SWI/SNF related, matrix associated, actin dependent regulator of chromatin, subfamily b, member 1 (INI1) confirmed by immunohistochemistry, or
    * Molecular confirmation of tumor-specific bi-allelic INI1 loss/mutation if INI1 immunohistochemistry is not available; note that molecular confirmation of tumor-specific bi-allelic INI1 loss/mutation is encouraged in cases where INI1 immunohistochemistry is equivocal
* Patients must have a Lansky or Karnofsky performance status score of ≥ 50, corresponding to Eastern Cooperative Oncology Group (ECOG) categories 0, 1 or 2; use Karnofsky for patients > 16 years of age and Lansky for patients ≤ 16 years of age; Note: Patients who are unable to walk because of paralysis, but who are up in a wheelchair, will be considered ambulatory for the purpose of assessing the performance score
* Patients must have fully recovered from the acute toxic effects of all prior chemotherapy, immunotherapy, or radiotherapy prior to study enrollment
* Myelosuppressive chemotherapy:

  * Solid tumors:

    * Patients with solid tumors must not have received myelosuppressive chemotherapy within 3 weeks of enrollment onto this study (6 weeks if prior nitrosourea)
  * Leukemia:

    * Patients with leukemia who relapse while receiving standard maintenance therapy will not be required to have a waiting period before enrollment onto this study
    * Patients who relapse while they are not receiving standard maintenance therapy must have completely recovered from all acute toxic effects of chemotherapy, immunotherapy or radiotherapy prior to study enrollment; at least 14 days must have elapsed since the completion of cytotoxic therapy, with the exception of hydroxyurea
    * Note: cytoreduction with hydroxyurea can be initiated and continued for up to 24 hours prior to the start of MLN8237
* At least 7 days must have elapsed since the completion of therapy with a growth factor; at least 14 days must have elapsed after receiving pegfilgrastim
* At least 7 days must have elapsed since completion of therapy with a biologic agent; for agents that have known adverse events occurring beyond 7 days after administration, this period prior to enrollment must be extended beyond the time during which adverse events are known to occur
* At least 3 half-lives must have elapsed since prior therapy that included a monoclonal antibody
* ≥ 2 weeks must have elapsed since local palliative radiation therapy (XRT) (small port); ≥ 6 weeks must have elapsed since treatment with therapeutic doses of MIBG; ≥ 6 months must have elapsed if prior craniospinal XRT was received, if ≥ 50% of the pelvis was irradiated, or if total body irradiation (TBI) was received; ≥ 6 weeks must have elapsed if other substantial bone marrow irradiation was given
* No evidence of active graft vs. host disease and ≥ 3 months must have elapsed since transplant
* For patients with solid tumors without bone marrow involvement:

  * Peripheral absolute neutrophil count (ANC) >= 1000/mm^3
  * Platelet count >= 100,000/mm^3 (transfusion independent, defined as not receiving platelet transfusions within a 7 day period prior to enrollment)
  * Hemoglobin > 8.0 g/dL (may receive red blood cell [RBC] transfusions)
* For patients with solid tumors and known bone marrow metastatic disease:

  * Peripheral absolute neutrophil count (ANC) ≥ 750/mm^3
  * Platelet count ≥ 50,000/mm^3
  * Hemoglobin ≥ 8.0 g/dL
  * Transfusions are permitted to meet both the platelet and hemoglobin criteria; patients must not be known to be refractory to red blood cell or platelet transfusions
* Patients with leukemia must not be known to be refractory to red blood cell or platelet transfusions
* Creatinine clearance or radioisotope glomerular filtration rate (GFR) 70 mL/min/1.73 m^2 or a serum creatinine based on age/gender as follows:

  * 1 to < 2 years: 0.6
  * 2 to < 6 years: 0.8
  * 6 to < 10 years: 1
  * 10 to < 13 years: 1.2
  * 13 to < 16 years: 1.5 (male), 1.4 (female)
  * >= 16 years: 1.7 (male), 1.4 (female)
* Total bilirubin =< 1.5 x upper limit of normal (ULN) for age
* Serum glutamic pyruvate transaminase (SGPT) (alanine aminotransferase [ALT]) ≤ 5.0 x ULN for age (≤ 225 U/L); for the purpose of this study, the ULN for SGPT is 45 U/L
* Serum albumin ≥ 2 g/dL
* All patients and/or their parents or legal guardians must sign a written informed consent

Exclusion Criteria:

* Patients who are pregnant or breast-feeding are not eligible for this study; negative pregnancy tests must be obtained in girls who are post-menarchal; males or females of reproductive potential may not participate unless they have agreed to use an effective contraceptive method for the duration of study therapy; breastfeeding women are excluded
* Growth factors that support platelet or white cell number or function must not have been administered within the 7 days prior to enrollment (14 days if pegfilgrastim)
* Patients requiring corticosteroids who have not been on a stable or decreasing dose of corticosteroid for the 7 days prior to enrollment are not eligible
* Patients who are currently receiving another investigational drug are not eligible
* Patients who are currently receiving other anti-cancer agents are not eligible
* Use of daily benzodiazepine therapy excludes a patient from being eligible because of the potential benzodiazepine-like effects of MLN8237
* Patients who are currently receiving digoxin, cyclosporine, tacrolimus, or sirolimus are not eligible
* Patients who are unable to swallow tablets are not eligible
* Patients who have an uncontrolled infection are not eligible
* Leukemia patients with CNS disease are not eligible
* Patients who in the opinion of the investigator may not be able to comply with the safety monitoring requirements of the study are not eligible

Ages: 1 Year to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 118 (Actual)
Dates: Start 2011-02; Primary Completion 2015-12-31 (Actual); Study Completion 2019-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yael Mosse, Principal Investigator — Children's Oncology Group
Locations (105):
- United States (97):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Southern California Permanente Medical Group, Downey, California
  - Miller Children's and Women's Hospital Long Beach, Long Beach, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Children's Hospital Central California, Madera, California
  - Children's Hospital of Orange County, Orange, California
  - Lucile Packard Children's Hospital Stanford University, Palo Alto, California
  - Rady Children's Hospital - San Diego, San Diego, California
  - UCSF Medical Center-Parnassus, San Francisco, California
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Yale University, New Haven, Connecticut
  - Alfred I duPont Hospital for Children, Wilmington, Delaware
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Lee Memorial Health System, Fort Myers, Florida
  - Nemours Children's Clinic-Jacksonville, Jacksonville, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Florida Hospital Orlando, Orlando, Florida
  - Nemours Children's Clinic - Orlando, Orlando, Florida
  - UF Cancer Center at Orlando Health, Orlando, Florida
  - Nemours Children's Clinic - Pensacola, Pensacola, Florida
  - All Children's Hospital, St. Petersburg, Florida
  - Saint Joseph's Hospital/Children's Hospital-Tampa, Tampa, Florida
  - Children's Healthcare of Atlanta - Egleston, Atlanta, Georgia
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Lurie Children's Hospital-Chicago, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Saint Jude Midwest Affiliate, Peoria, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Riley Hospital for Children, Indianapolis, Indiana
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Tulane University Health Sciences Center, New Orleans, Louisiana
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Children's Hospitals and Clinics of Minnesota - Minneapolis, Minneapolis, Minnesota
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - The Childrens Mercy Hospital, Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Children's Hospital and Medical Center of Omaha, Omaha, Nebraska
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Rutgers Cancer Institute of New Jersey-Robert Wood Johnson University Hospital, New Brunswick, New Jersey
  - Overlook Hospital, Summit, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Roswell Park Cancer Institute, Buffalo, New York
  - Winthrop University Hospital, Mineola, New York
  - Columbia University/Herbert Irving Cancer Center, New York, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - New York Medical College, Valhalla, New York
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Novant Health Presbyterian Medical Center, Charlotte, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Rainbow Babies and Childrens Hospital, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Dayton Children's Hospital, Dayton, Ohio
  - Mercy Children's Hospital, Toledo, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Natalie Warren Bryant Cancer Center at Saint Francis, Tulsa, Oklahoma
  - Legacy Emanuel Children's Hospital, Portland, Oregon
  - Legacy Emanuel Hospital and Health Center, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Penn State Hershey Children's Hospital, Hershey, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Childrens Oncology Group, Philadelphia, Pennsylvania
  - Saint Christopher's Hospital for Children, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Palmetto Health Richland, Columbia, South Carolina
  - East Tennessee Childrens Hospital, Knoxville, Tennessee
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Driscoll Children's Hospital, Corpus Christi, Texas
  - Medical City Dallas Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - Methodist Children's Hospital of South Texas, San Antonio, Texas
  - University of Vermont College of Medicine, Burlington, Vermont
  - Childrens Hospital-King's Daughters, Norfolk, Virginia
  - Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia
  - Carilion Clinic Children's Hospital, Roanoke, Virginia
  - Seattle Children's Hospital, Seattle, Washington
  - Providence Sacred Heart Medical Center and Children's Hospital, Spokane, Washington
  - Saint Vincent Hospital, Green Bay, Wisconsin
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
  - Children¿s Hospital of Wisconsin, Milwaukee, Wisconsin
- Canada (8):
  - Alberta Children's Hospital, Calgary, Alberta
  - British Columbia Children's Hospital, Vancouver, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - IWK Health Centre, Halifax, Nova Scotia
  - Cancer Centre of Southeastern Ontario at Kingston General Hospital, Kingston, Ontario
  - Hospital for Sick Children, Toronto, Ontario
  - The Montreal Children's Hospital of the MUHC, Montreal, Quebec
  - Centre Hospitalier Universitaire Sainte-Justine, Montreal, Quebec

REFERENCES:
- [Derived] Zhou X, Mould DR, Yuan Y, Fox E, Greengard E, Faller DV, Venkatakrishnan K. Population Pharmacokinetics and Exposure-Safety Relationships of Alisertib in Children and Adolescents With Advanced Malignancies. J Clin Pharmacol. 2022 Feb;62(2):206-219. doi: 10.1002/jcph.1958. Epub 2022 Jan 15. PMID 34435684
- [Derived] Mosse YP, Fox E, Teachey DT, Reid JM, Safgren SL, Carol H, Lock RB, Houghton PJ, Smith MA, Hall D, Barkauskas DA, Krailo M, Voss SD, Berg SL, Blaney SM, Weigel BJ. A Phase II Study of Alisertib in Children with Recurrent/Refractory Solid Tumors or Leukemia: Children's Oncology Group Phase I and Pilot Consortium (ADVL0921). Clin Cancer Res. 2019 Jun 1;25(11):3229-3238. doi: 10.1158/1078-0432.CCR-18-2675. Epub 2019 Feb 18. PMID 30777875

RESULTS

PARTICIPANT FLOW:
Groups:
- Recurrent Neuroblastoma With Measurable Disease at Enrollment: Experimental: Arm 1
- Recurrent Neuroblastoma Only MIBG Evaluable Disease at Enroll: Experimental: Arm 2
- Previously Treated Childhood Rhabdomyosarcoma: Experimental: Arm 3
- Recurrent Osteosarcoma: Experimental: Arm 4
- Recurrent Ewing Sarcoma /Peripheral Neuroectodermal Tumor: Experimental: Arm 5
- Recurrent Childhood Soft Tissue Sarcoma: Experimental: Arm 6
- Childhood Hepatoblastoma: Experimental: Arm 7
- Recurrent Childhood Germ Cell Tumor: Experimental: Arm 8
- Recurrent Wilms Tumor and Other Childhood Kidney Tumors: Experimental: Arm 9
- Recurrent Childhood Acute Lympohblastic Leukemia: Experimental: Arm 10
- Recurrent Childhood Acute Myeloid Leukemia: Experimental: Arm 11
- Rhaboid Malignancy: Experimental: Arm 12
Period: Overall Study
Arm/Group | Recurrent Neuroblastoma With Measurable Disease at Enrollment | Recurrent Neuroblastoma Only MIBG Evaluable Disease at Enroll | Previously Treated Childhood Rhabdomyosarcoma | Recurrent Osteosarcoma | Recurrent Ewing Sarcoma /Peripheral Neuroectodermal Tumor | Recurrent Childhood Soft Tissue Sarcoma | Childhood Hepatoblastoma | Recurrent Childhood Germ Cell Tumor | Recurrent Wilms Tumor and Other Childhood Kidney Tumors | Recurrent Childhood Acute Lympohblastic Leukemia | Recurrent Childhood Acute Myeloid Leukemia | Rhaboid Malignancy
Started | 20 | 12 | 10 | 10 | 10 | 8 | 6 | 7 | 10 | 10 | 11 | 4
Completed | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not Completed | 20 | 10 | 10 | 10 | 10 | 8 | 6 | 7 | 9 | 10 | 11 | 4
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 3 | 0 | 0
Not completed — Progressive Disease | 13 | 8 | 9 | 9 | 8 | 8 | 5 | 6 | 8 | 6 | 10 | 3
Not completed — Physician Decision | 1 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Not completed — Adverse Event | 5 | 2 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Recurrent Neuroblastoma With Measurable Disease at Enrollment | Recurrent Neuroblastoma Only MIBG Evaluable Disease at Enroll | Previously Treated Childhood Rhabdomyosarcoma | Recurrent Osteosarcoma | Recurrent Ewing Sarcoma /Peripheral Neuroectodermal Tumor | Recurrent Childhood Soft Tissue Sarcoma | Childhood Hepatoblastoma | Recurrent Childhood Germ Cell Tumor | Recurrent Wilms Tumor and Other Childhood Kidney Tumors | Recurrent Childhood Acute Lympohblastic Leukemia | Recurrent Childhood Acute Myeloid Leukemia | Rhaboid Malignancy | Total
Number analyzed (Participants) | 20 | 12 | 10 | 10 | 10 | 8 | 6 | 7 | 10 | 10 | 11 | 4 | 118
Age, Continuous [Median (Full Range); unit: Years] | 8 [3 to 20] | 8 [5 to 17] | 12 [4 to 21] | 17 [12 to 21] | 14 [6 to 20] | 16 [13 to 21] | 5 [3 to 14] | 11 [3 to 19] | 10 [3 to 18] | 13 [7 to 19] | 10 [3 to 15] | 5 [2 to 7] | 11 [2 to 21]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 2 | 7 | 3 | 3 | 4 | 1 | 4 | 7 | 3 | 6 | 2 | 52
  Male | 10 | 10 | 3 | 7 | 7 | 4 | 5 | 3 | 3 | 7 | 5 | 2 | 66
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 1 | 1 | 3 | 1 | 2 | 3 | 2 | 4 | 2 | 4 | 1 | 27
  Not Hispanic or Latino | 15 | 10 | 7 | 7 | 8 | 5 | 3 | 4 | 5 | 8 | 5 | 3 | 80
  Unknown or Not Reported | 2 | 1 | 2 | 0 | 1 | 1 | 0 | 1 | 1 | 0 | 2 | 0 | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 1 | 1 | 2 | 0 | 1 | 1 | 0 | 2 | 2 | 2 | 0 | 14
  White | 15 | 7 | 7 | 7 | 8 | 3 | 3 | 4 | 5 | 5 | 2 | 3 | 69
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 3 | 4 | 2 | 1 | 2 | 4 | 2 | 3 | 3 | 3 | 7 | 1 | 35
Region of Enrollment [Number; unit: participants] — Region unknown for 1 patient in the Recurrent Wilms Tumor and Other Childhood Kidney Tumors arm.
  participants
    Canada | 1 | 2 | 1 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 0 | 8
    United States | 18 | 9 | 9 | 10 | 10 | 8 | 5 | 6 | 8 | 10 | 10 | 4 | 107
    United Kingdom | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Overall Response
Description: For patients with recurrent solid tumors a patient who experienced a complete or partial response according to RECIST version 1.1 criteria is considered a responder. For patients with recurrent acute lymphoblastic leukemia a patient who experiences a bone marrow evaluation with < 5% blast cells on morphological evaluation of bone marrow will be considered a responder. For patients with recurrent acute myelogenous leukemia a patient who experiences a complete remission or complete remission with partial recovery of platelet count according to the AML International Working Group Criteria will be considered a responder.
Time Frame: From first dose of alisertib through 6 cycles of protocol therapy or until removal from protocol therapy whichever occurred first.
Population: Of the 118 enrolled patients, two were not evaluable for the primary outcome measure. Neither received protocol therapy. One was enrolled in arm 11, one was enrolled in Arm 1.
Measure: Number; unit: Patients
Arm/Group | Recurrent Neuroblastoma With Measurable Disease at Enrollment | Recurrent Neuroblastoma Only MIBG Evaluable Disease at Enroll | Previously Treated Childhood Rhabdomyosarcoma | Recurrent Osteosarcoma | Recurrent Ewing Sarcoma /Peripheral Neuroectodermal Tumor | Recurrent Childhood Soft Tissue Sarcoma | Childhood Hepatoblastoma | Recurrent Childhood Germ Cell Tumor | Recurrent Wilms Tumor and Other Childhood Kidney Tumors | Recurrent Childhood Acute Lympohblastic Leukemia | Recurrent Childhood Acute Myeloid Leukemia | Rhaboid Malignancy
Number analyzed (Participants) | 19 | 12 | 10 | 10 | 10 | 8 | 6 | 7 | 10 | 10 | 10 | 4
Patients | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0

2. Secondary Outcome: Number of Patients Cycles With Grade 3 or Higher Adverse Event
Description: The number of patient-cycles in which the adverse event considered grade 3 or higher AE according to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 considered by the treating physician to be possibly, probably or definitely related to alisertib.
Time Frame: Up to 24 months
Population: 116 patients contributed 360 patient-cycles to the analysis.
Measure: Number; unit: Patient-cycle
Groups:
- All Patients: All patients
Arm/Group | All Patients
Number analyzed (Participants) | 116
Patient-cycle
  Abdominal Pain | 3
  Prolonged Partial Thromboplatin Time | 1
  Acute Kidney Injury | 1
  Agitation | 1
  Alanine Aminotransferase Elevation | 25
  Allergic Reaction | 1
  Alopecia | 27
  Anal Mucocitis | 1
  Anemia | 141
  Anorexia | 8
  Aspartate Aminotransferase Increase | 15
  Back Pain | 1
  Blood Bilirubin Increase | 7
  Blurred Vision | 2
  Bullous Dermatitis | 1
  Colitis | 2
  Confusion | 1
  Dehydration | 5
  Depression | 1
  Diarrhea | 8
  Dizziness | 15
  Dry Mouth | 1
  Enterocolitis | 1
  Erectile Dysfunction | 1
  Euphoria | 3
  Eye Pain | 1
  Fatigue | 14
  Febrile Neutropenia | 13
  Other Gastrointestinal Disorders | 1
  GGT Increase | 2
  Headache | 3
  Hepatic Hemhorrage | 1
  Hyperkalemia | 1
  Hypersomnia | 1
  Hyperuricemia | 1
  Hypoalbuminemia | 7
  Hypocalcemia | 2
  Hypokalemia | 9
  Hyponatremia | 3
  Hypophosphatemia | 1
  Other Infections | 1
  INR Increase | 1
  Keratitis | 1
  Lethargy | 1
  Lung Infection | 1
  Lymphocyte Count Decrease | 65
  Lymphocyte Count Increase | 1
  Mucosal Infection | 2
  Oral Mucocitis | 35
  Nausea | 11
  Decreased Neutrophil Count | 208
  Oral Pain | 12
  Otitis Media | 1
  Pain in an Extremity | 1
  Palmar-Plantar Erythrodysesthesia Syndrome | 10
  Photophobia | 4
  Platelet Count Decrease | 92
  Pruritis | 4
  Psychiatric Disorders | 1
  Respiratory Failure | 1
  Serum Amylase Increase | 1
  Skin Infection | 1
  Somnolence | 2
  Sore Throat | 1
  Tumor Lysis Syndrome | 1
  Upper Respiratory Infection | 1
  Urticaria | 1
  Urinary Tract Infection | 4
  Vomiting | 1
  White Blood Cell Decrease | 163

3. Secondary Outcome: Serum Concentration of Alisertib Prior to the First Day of Administration
Description: Serum concentration of alisertib prior to the first day of administration in nanograms/milliliter.
Time Frame: day 1 of protocol therapy
Population: Of all eligible patients enrolled, 32 provided a prior to the first day of administration sample for analysis.
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | All Patients
Number analyzed (Participants) | 32
ng/ml | 0 (0)

4. Secondary Outcome: Serum Concentration of Alisertib on the First Day of Administration One Hour After Administration
Description: Serum concentration of alisertib on the first day of administration one hour after administration in nanograms/milliliter.
Time Frame: day 1 of protocol therapy
Population: Of all eligible patients enrolled, 16 provided a first day of administration one hour after administration infusion sample for analysis.
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | All Patients
Number analyzed (Participants) | 16
ng/ml | 1874.0625 (1131.87375)

5. Secondary Outcome: Serum Concentration of Alisertib on the First Day of Administration Three Hours After Administration
Description: Serum concentration of alisertib on the first day of administration three hours after administration in nanograms/milliliter.
Time Frame: day 1 of protocol therapy
Population: Of all eligible patients enrolled, 16 provided a first day of administration three hours after administration sample for analysis.
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | All Patients
Number analyzed (Participants) | 16
ng/ml | 1863.9375 (588.116822)

6. Secondary Outcome: Serum Concentration of Alisertib on the First Day of Administration Six Hours After Administration
Description: Serum concentration of alisertib on the first day of administration six hours after administration in nanograms/milliliter.
Time Frame: day 1 of protocol therapy
Population: Of all eligible patients enrolled, 16 provided a first day of administration six hours after administration sample for analysis.
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | All Patients
Number analyzed (Participants) | 16
ng/ml | 1234 (512.203475)

7. Secondary Outcome: Serum Concentration of Alisertib on the Fourth Day of Administration Prior to the Administration of the Day 4 Dose
Description: Serum concentration of alisertib on the fourth day of administration prior to the administration of the day 4 dose in nanograms/milliliter.
Time Frame: day 4 of protocol therapy
Population: Of all eligible patients enrolled, 30 provided a fourth day of administration prior to the administration of the day 4 dose sample for analysis.
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | All Patients
Number analyzed (Participants) | 30
ng/ml | 1123.73333 (715.013235)

8. Secondary Outcome: Serum Concentration of Alisertib on the Seventh Day of Administration Prior to the Administration of the Day 7 Dose.
Description: Serum concentration of alisertib on the seventh day of administration prior to the administration of the day 7 dose in nanograms/milliliter.
Time Frame: day 7 of protocol therapy
Population: Of all eligible patients enrolled, 31 provided a seventh day of administration prior to the administration of the day 7 dose sample for analysis.
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | All Patients
Number analyzed (Participants) | 31
ng/ml | 1097.50645 (1012.34016)

ADVERSE EVENTS:
Groups:
- Rhaboid Malignancy: Experimental: 12
Arm/Group | Recurrent Neuroblastoma With Measurable Disease at Enrollment | Recurrent Neuroblastoma Only MIBG Evaluable Disease at Enroll | Previously Treated Childhood Rhabdomyosarcoma | Recurrent Osteosarcoma | Recurrent Ewing Sarcoma /Peripheral Neuroectodermal Tumor | Recurrent Childhood Soft Tissue Sarcoma | Childhood Hepatoblastoma | Recurrent Childhood Germ Cell Tumor | Recurrent Wilms Tumor and Other Childhood Kidney Tumors | Recurrent Childhood Acute Lympohblastic Leukemia | Recurrent Childhood Acute Myeloid Leukemia | Rhaboid Malignancy
Serious Adverse Events (participants affected / at risk) | 7/20 | 5/12 | 4/10 | 7/10 | 5/10 | 3/8 | 6/6 | 1/7 | 3/10 | 8/10 | 5/11 | 2/4
Other Adverse Events (participants affected / at risk) | 15/20 | 11/12 | 8/10 | 9/10 | 9/10 | 6/8 | 3/6 | 5/7 | 9/10 | 10/10 | 9/11 | 2/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Recurrent Neuroblastoma With Measurable Disease at Enrollment (N=20) | Recurrent Neuroblastoma Only MIBG Evaluable Disease at Enroll (N=12) | Previously Treated Childhood Rhabdomyosarcoma (N=10) | Recurrent Osteosarcoma (N=10) | Recurrent Ewing Sarcoma /Peripheral Neuroectodermal Tumor (N=10) | Recurrent Childhood Soft Tissue Sarcoma (N=8) | Childhood Hepatoblastoma (N=6) | Recurrent Childhood Germ Cell Tumor (N=7) | Recurrent Wilms Tumor and Other Childhood Kidney Tumors (N=10) | Recurrent Childhood Acute Lympohblastic Leukemia (N=10) | Recurrent Childhood Acute Myeloid Leukemia (N=11) | Rhaboid Malignancy (N=4)
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Activated partial thromboplastin time prolonged (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Agitation (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Allergic reaction (Immune system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Anorectal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cardiac disorders - Other, specify (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Catheter related infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Colitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Death NOS (General disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Enterocolitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Enterocolitis infectious (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 5 | 4 | 0
Fever (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hematoma (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hepatic hemorrhage (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypersomnia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperuricemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 3 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Hypocalcemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Hypoglycemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypokalemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 1
Hyponatremia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Infections and infestations - Other, specify (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
INR increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Intracranial hemorrhage (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Keratitis (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lung infection (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Lymphocyte count decreased (Investigations) | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Mucositis oral (Gastrointestinal disorders) | 3 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Myositis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Platelet count decreased (Investigations) | 1 | 1 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Seizure (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tumor lysis syndrome (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper respiratory infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urine output decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
White blood cell decreased (Investigations) | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Recurrent Neuroblastoma With Measurable Disease at Enrollment (N=20) | Recurrent Neuroblastoma Only MIBG Evaluable Disease at Enroll (N=12) | Previously Treated Childhood Rhabdomyosarcoma (N=10) | Recurrent Osteosarcoma (N=10) | Recurrent Ewing Sarcoma /Peripheral Neuroectodermal Tumor (N=10) | Recurrent Childhood Soft Tissue Sarcoma (N=8) | Childhood Hepatoblastoma (N=6) | Recurrent Childhood Germ Cell Tumor (N=7) | Recurrent Wilms Tumor and Other Childhood Kidney Tumors (N=10) | Recurrent Childhood Acute Lympohblastic Leukemia (N=10) | Recurrent Childhood Acute Myeloid Leukemia (N=11) | Rhaboid Malignancy (N=4)
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1
Activated partial thromboplastin time prolonged (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 4 | 3 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 2 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 6 | 1 | 2 | 1 | 3 | 0 | 0 | 2 | 0 | 0 | 0 | 1
Anal mucositis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anemia (Blood and lymphatic system disorders) | 9 | 7 | 5 | 5 | 3 | 1 | 2 | 1 | 6 | 7 | 7 | 2
Anorexia (Metabolism and nutrition disorders) | 2 | 1 | 0 | 2 | 3 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 3 | 2 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 2 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 1 | 2 | 2 | 0
Blurred vision (Eye disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bullous dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Catheter related infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chills (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Concentration impairment (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Confusion (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Creatinine increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Diarrhea (Gastrointestinal disorders) | 3 | 1 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Enterocolitis infectious (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Euphoria (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Eye pain (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Fatigue (General disorders) | 3 | 1 | 1 | 2 | 3 | 0 | 0 | 0 | 1 | 0 | 1 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 1 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Fever (General disorders) | 0 | 3 | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gait disturbance (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
GGT increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0
Headache (Nervous system disorders) | 1 | 1 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1
Hearing impaired (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypercalcemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Hypermagnesemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0
Hypocalcemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 2 | 1 | 0
Hypokalemia (Metabolism and nutrition disorders) | 1 | 1 | 2 | 1 | 1 | 0 | 1 | 0 | 0 | 4 | 0 | 0
Hyponatremia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Hypophosphatemia (Metabolism and nutrition disorders) | 1 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 2 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Infections and infestations - Other, specify (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Injury, poisoning and procedural complications - Other, specify (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
INR increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lethargy (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lymphocyte count decreased (Investigations) | 10 | 4 | 3 | 5 | 5 | 3 | 1 | 1 | 2 | 4 | 4 | 0
Lymphocyte count increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Mucosal infection (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mucositis oral (Gastrointestinal disorders) | 3 | 4 | 3 | 1 | 3 | 1 | 1 | 1 | 2 | 1 | 3 | 0
Nausea (Gastrointestinal disorders) | 3 | 0 | 2 | 2 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Neutrophil count decreased (Investigations) | 15 | 10 | 6 | 7 | 4 | 1 | 2 | 4 | 7 | 2 | 6 | 2
Oral pain (Gastrointestinal disorders) | 0 | 1 | 2 | 1 | 1 | 0 | 0 | 1 | 1 | 1 | 0 | 0
Otitis media (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pain (General disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 2 | 1 | 0 | 0 | 1 | 0 | 2 | 0 | 0
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 | 2 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Peripheral motor neuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Photophobia (Eye disorders) | 0 | 1 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Platelet count decreased (Investigations) | 11 | 5 | 4 | 4 | 3 | 1 | 2 | 2 | 5 | 7 | 6 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Proteinuria (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Psychiatric disorders - Other, specify (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Scrotal infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Seizure (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Serum amylase increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Testicular hemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper respiratory infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 1 | 0 | 1 | 0 | 1 | 0 | 1 | 2 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Weight gain (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Weight loss (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
White blood cell decreased (Investigations) | 13 | 8 | 5 | 7 | 7 | 0 | 2 | 4 | 6 | 4 | 4 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Must obtain prior Sponsor approval.